CLINICAL TRIAL: NCT00923091
Title: Randomised, Double-Blind, Parallel-Group Study Evaluating Efficacy and Safety of Co-Administration of Triple Combinations of Olmesartan Medoxomil, Amlodipine Besylate, and Hydrochlorothiazide Compared With Corresponding Olmesartan - Amlodipine Combination in Subjects With Hypertension
Brief Title: Parallel-Group Comparison of Olmesartan (OLM), Amlodipine (AML) and Hydrochlorothiazid (HCTZ) in Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS8635-A-E302
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2012-04

CONDITIONS: Essential Hypertension
Keywords: triple combination; parallel group; dual combination
MeSH Terms: conditions — Essential Hypertension | interventions — Olmesartan Medoxomil; Amlodipine; Amlodipine Besylate, Olmesartan Medoxomil Drug Combination; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- olmesartan/amlodipine/hydrochlorothiazide 20mg/5mg/12.5mg (Experimental): olmesartan medoxomil 20mg / amlodipine besylate 5 mg / hydrochlorothiazide 12.5mg
  Interventions: Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide + placebo
- olmesartan/amlodipine/hydrochlorothiazide 40mg/5mg/12.5mg (Experimental)
  Interventions: Drug: Olmesartan medoxomil + amlodipine + hydrochlorothiazide + placebo
- olmesartan/amlodipine/hydrochlorothiazide 40mg/5mg/25mg (Experimental)
  Interventions: Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide
- olmesartan/amlodipine/hydrochlorothiazide 40mg/10mg/12.5mg (Experimental)
  Interventions: Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide
- olmesartan/amlodipine/hydrochlorothiazide 40mg/10mg/25mg (Experimental)
  Interventions: Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide
- olmesartan/amlodipine 20mg/5mg (Experimental): olmesartan medoxomil 20mg / amlodipine besylate 5mg
  Interventions: Drug: olmesartan medoxomil + amlodipine
- olmesartan/amlodipine 40mg/5mg (Experimental)
  Interventions: Drug: olmesartan medoxomil + amlodipine
- olmesartan/amlodipine 40mg/10mg (Experimental)
  Interventions: Drug: olmesartan medoxomil + amlodipine

INTERVENTIONS:
Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide + placebo — One olmesartan medoxomil 20 mg + amlodipine 5 mg combination oral tablet taken once per day. One hydrochlorothiazide 12.5 mg tablet + one hydrochlorothiazide 12.5 mg placebo tablet taken once per day.
  Other Names: Azor
  Arms: olmesartan/amlodipine/hydrochlorothiazide 20mg/5mg/12.5mg
Drug: Olmesartan medoxomil + amlodipine + hydrochlorothiazide + placebo — One olmesartan medoxomil 40 mg + amlodipine 5 mg combination oral tablet taken once per day. One hydrochlorothiazide 12.5 mg tablet + one hydrochlorothiazide 12.5 mg placebo tablet taken once per day.
  Other Names: Azor
  Arms: olmesartan/amlodipine/hydrochlorothiazide 40mg/5mg/12.5mg
Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide — One olmesartan medoxomil 40 mg + amlodipine 5 mg combination oral tablet taken once per day. Two hydrochlorothiazide 12.5 mg tablets taken once per day.
  Other Names: Azor; Norvasc
  Arms: olmesartan/amlodipine/hydrochlorothiazide 40mg/5mg/25mg
Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide — One olmesartan medoxomil 40 mg + amlodipine 10 mg combination oral tablet taken once per day. One hydrochlorothiazide 12.5 mg tablet + one hydrochlorothiazide 12.5 mg placebo tablet taken once per day.
  Other Names: Azor
  Arms: olmesartan/amlodipine/hydrochlorothiazide 40mg/10mg/12.5mg
Drug: olmesartan medoxomil + amlodipine + hydroclororthiazide — One olmesartan medoxomil 40 mg + amlodipine 10 mg combination oral tablet taken once per day. Two hydrochlorothiazide 12.5 mg tablets taken once per day.
  Other Names: Azor
  Arms: olmesartan/amlodipine/hydrochlorothiazide 40mg/10mg/25mg
Drug: olmesartan medoxomil + amlodipine — One olmesartan medoxomil 20 mg + amlodipine 5 mg combination oral tablet taken once per day
  Other Names: Azor
  Arms: olmesartan/amlodipine 20mg/5mg
Drug: olmesartan medoxomil + amlodipine — One olmesartan medoxomil 40 mg + amlodipine 5 mg combination oral tablet taken once per day.
  Arms: olmesartan/amlodipine 40mg/5mg
Drug: olmesartan medoxomil + amlodipine — One olmesartan medoxomil 40 mg + amlodipine 10 mg combination oral tablet taken once per day.
  Other Names: Azor
  Arms: olmesartan/amlodipine 40mg/10mg

SUMMARY:
This study is to determine the change in blood pressure from the administration of Olmesartan/Amlodipine/Hydrochlorothiazide triple combinations compared to dual combinations with Olmesartan/Amlodipine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older.
* Subjects with mean trough seated blood pressure (SeBP) ≥ 160/100 mmHg, (seated systolic blood pressure(SeSBP) ≥ 160 mmHg and seated diastolic blood pressure (SeDBP) ≥ 100 mmHg) at Screening if not currently on antihypertensive medication (newly diagnosed subjects or subjects who are not taking any antihypertensive medication for at least 3 weeks); Or Subjects with mean trough SeBP ≥ 160/100 mmHg, SeSBP ≥ 160 mmHg and SeDBP ≥ 100 mmHg) after washout of prior antihypertensive medication in subjects who discontinued their previous antihypertensive medication.

The difference in mean SeSBP/SeDBP between the visit prior to randomisation and the randomisation visit must be ≤ 20/10 mmHg. Subjects not currently on antihypertensive (HTN) medication may meet this requirement at the screening visit (Visit 1) and the randomization visit (Visit 3). Subjects washing out of HTN medication must meet this requirement at least by Visit 2 (or Visit 2.1, if needed) and Visit 3. All subjects undergoing washout of their prior antihypertensive medication will have the opportunity to re-visit the study sites for additional visits during washout (Visits 2 and 2.1) to assess eligibility for randomisation.

* Subjects freely sign the informed consent form (ICF) after the nature of the study and the disclosure of his/her data has been explained.
* Female subjects of childbearing potential must be using adequate contraception (female of childbearing potential is defined as one who has not been postmenopausal for at least one year, or has not been surgically sterilised, or has not had a hysterectomy at least three months prior to the start of this study [Visit 1]). Adequate contraceptives include hormonal intra-uterine devices, hormonal contraceptives (oral, depot, patch or injectable), and double barrier methods such as condoms or diaphragms with spermicidal gel or foam.

Exclusion Criteria:

* Female subjects of childbearing potential who are pregnant or lactating.
* Subjects with serious disorders which may limit the ability to evaluate the efficacy or safety of the investigational products, including cerebrovascular, cardiovascular, renal, respiratory, hepatic, gastrointestinal, endocrine or metabolic, haematologic or, neurologic, and psychiatric diseases. The same applies for immunocompromised and/or neutropenic subjects.
* Subjects having a history of the following within the last six months: myocardial infarction (MI), unstable angina pectoris, percutaneous coronary intervention, heart failure, hypertensive encephalopathy, cerebrovascular accident (stroke), or transient ischaemic attack.
* Subjects with clinically significant abnormal laboratory values at Screening, including subjects with one or more of the following:

  * Aspartate aminotransferase (AST) > 3 times upper limit of normal (ULN).
  * Alanine aminotransferase (ALT) > 3 times ULN.
  * Gamma-glutamyl transferase (GGT) > 3 times ULN.
  * Potassium above ULN (unless high value is due to haemolytic blood sample).
* Subjects with secondary hypertension of any aetiology such as renal disease, phaeochromocytoma, or Cushing's syndrome.
* Subjects with contraindication to olmesartan, amlodipine, hydrochlorothiazide, or any of the tablet's excipients.
* Newly diagnosed subjects with a mean trough SeSBP > 200 mmHg or mean trough SeDBP > 115 mmHg or any subjects with bradycardia (heart rate < 50 beats/min at rest documented by mean radial pulse rate [PR] or electrocardiogram [ECG]) at Screening (Visit 1) or immediately before taking Period I study medication (Visit 3).
* Subjects already taking four or more antihypertensive medications.
* Subjects with a mean trough SeSBP > 145 mmHg or mean trough SeDBP > 95 mmHg while taking three antihypertensive medications.
* Subjects with a mean trough SeSBP > 160 mmHg or mean trough SeDBP > 100 mmHg while taking two antihypertensive medications.
* Subjects with a mean trough SeSBP > 180 mmHg or mean trough SeDBP > 110 mmHg while taking one antihypertensive medication.
* Subjects with electrocardiogram evidence of 2nd or 3rd degree atrio ventricular (AV) block, atrial fibrillation, or other cardiac arrhythmia (requiring treatment).
* Subjects with severe heart failure (New York Heart Association stage III-IV), clinically significant aortic or mitral valve stenosis, uncorrected coarctation of the aorta, obstruction of cardiac outflow (obstructive, hypertrophic cardiomyopathy) or symptomatic coronary disease.
* Subjects with clinical evidence of renal disease including reno-vascular occlusive disease, nephrectomy and/or renal transplant, bilateral renal artery stenosis, unilateral renal artery stenosis in a solitary kidney, or severe renal impairment as evidenced by CrCl of < 30 mL/min calculated using the Cockcroft and Gault formula.
* Subjects with clinically relevant hepatic impairment.
* Subjects with biliary obstruction.
* Subjects with uncontrolled Type 1 or Type 2 diabetes defined as HbA1c > 9.0%. Diabetics must have documentation of HbA1c within 6 months of the Screening Visit, or must have their HbA1c assessed prior to randomisation. Note: subjects with Type 1 or Type 2 diabetes controlled with insulin, diet or oral hypoglycaemic agents on a stable dose for at least 30 days may be included.
* Subjects with a history of a wasting disease (e.g. cancer), autoimmune diseases, connective tissue diseases, major allergies or angioneurotic oedema.
* Subjects who require or are taking any concomitant medication which may interfere with the objectives of the study.
* Subjects on beta blockers or calcium channel blockers (CCBs) for both hypertension and either ischemia, post-MI prophylaxis or tachyarrhythmias.
* Subjects with known malabsorption syndromes.
* Subjects with psychiatric or emotional problems, which would invalidate the giving of informed consent or limit the ability of the subject to comply with study requirements.
* Subjects with a history of alcohol and/or drug abuse.
* Subjects who have received any investigational agent within 30 days prior to Screening.
* Subjects who are unwilling or unable to provide informed consent or to participate satisfactorily for the entire study.
* Subjects with malignancy during the past 2 years excluding squamous cell or basal cell carcinoma of the skin.
* Subjects with signs or symptoms which could exacerbate the occurrence of hypotension such as volume and salt depletion.
* Subjects with any medical condition, which in the judgment of the Investigator would jeopardise the evaluation of efficacy or safety and/or constitute a significant safety risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2689 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (133):
- Belgium (10):
  - Antwerp
  - Buizingen
  - De Pinte
  - Drongen
  - Ghent
  - Gilly
  - Merksem
  - Mouscron
  - Tremelo
  - Wichelen
- Bulgaria (6):
  - Burgas
  - Pleven
  - Plovdiv
  - Sofia
  - Stara Zagora
  - Veliko Tarnovo
- Czechia (10):
  - Benátky nad Jizerou
  - Brodce
  - Havířov
  - Jičín
  - Mladá Boleslav
  - Moravská Ostrava
  - Pilsen
  - Prachatice
  - Prague
  - Sokolov
- Denmark (3):
  - Copenhagen
  - Frederiksberg
  - Roskilde
- Germany (13):
  - Berlin
  - Cloppenburg
  - Delitzsch
  - Dresden
  - Erfurt
  - Essen
  - Hamburg
  - Heidelberg
  - Leipzig
  - Northeim
  - Simmern
  - Wallerfing
  - Wiesbaden
- Hungary (11):
  - Budapest
  - Debrecen
  - Hódmezővásárhely
  - Jászberény
  - Kaposvár
  - Kecskemét
  - Orosháza
  - Pécs
  - Székesfehérvár
  - Veszprém
  - Zalaegerszeg
- Italy (13):
  - Bologna
  - Brescia
  - Chieti
  - Ferrara
  - Foggia
  - Genova
  - Palermo
  - Parma
  - Perugia
  - Pisa
  - Roma
  - Sassari
  - Stradella Pavia
- Latvia (8):
  - Cēsis
  - Daugavpils
  - Jēkabpils
  - Ogre
  - Riga
  - Tukums
  - Varakļāni
  - Ventspils
- Netherlands (6):
  - Deurne
  - Eindhoven
  - Lichtenvoorde
  - Lieshout
  - Rotterdam
  - Utrecht
- Poland (12):
  - Bialystok
  - Dębica
  - Gdansk
  - Gdynia
  - Jastrzebia Zdroj
  - Krakow
  - Lublin
  - Mielec
  - Opole
  - Szczecin
  - Warsaw
  - Wroclaw
- Romania (9):
  - Arad
  - Bucharest
  - Craiova
  - Iași
  - Piteşti
  - Ploieşti
  - Sibiu
  - Suceava
  - Timișoara
- Russia (6):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tyumen
  - Yaroslavl
- Slovakia (6):
  - Banska Bysterica
  - Bratilslava
  - Nitra
  - Považská Bystrica
  - Rimavská Sobota
  - Žilina
- Spain (9):
  - Badalona
  - Barcelona
  - Ferrol
  - Lleida
  - Madrid
  - Petrel
  - Salamanca
  - Santiago de Compostela
  - Valencia
- Ukraine (11):
  - Dnipropetrovsk
  - Donetsk
  - Kharkiv
  - Kyiv
  - Lutsk
  - Lviv
  - Odesa
  - Simferopol
  - Vinnytsia
  - Zaporizhzhya
  - Zhytomyr

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Marques da Silva P, Haag U, Guest JF, Brazier JE, Soro M. Health-related quality of life impact of a triple combination of olmesartan medoxomil, amlodipine besylate and hydrochlorotiazide in subjects with hypertension. Health Qual Life Outcomes. 2015 Feb 21;13:24. doi: 10.1186/s12955-015-0216-6. PMID 25879524
- [Derived] Volpe M, de la Sierra A, Ammentorp B, Laeis P. Open-label study assessing the long-term efficacy and safety of triple olmesartan/amlodipine/hydrochlorothiazide combination therapy for hypertension. Adv Ther. 2014 May;31(5):561-74. doi: 10.1007/s12325-014-0117-9. Epub 2014 Apr 24. PMID 24760656
- [Derived] Volpe M, Christian Rump L, Ammentorp B, Laeis P. Efficacy and safety of triple antihypertensive therapy with the olmesartan/amlodipine/hydrochlorothiazide combination. Clin Drug Investig. 2012 Oct 1;32(10):649-64. doi: 10.1007/BF03261919. PMID 22909147

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conduct in Europe from 27 May 2009 to 12 January 2011
Pre-assignment Details: Study has randomised, double-blind, placebo-controlled parallel-group portion (Periods I-II) followed by transition phase (Periods III-V) wherein combination titration steps were evaluated in subjects not achieving blood pressure goals. The transition required that all be entered into Period 3 on olm/aml/hctz 20/5/12.5 to ensure a common baseline.
Groups:
- Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 20 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion. In Period III, all participants were included in this group. Responders (a participant was considered a responder if their blood pressure was <140/90 mm Hg; <130/80 mm Hg if the participant had diabetes or chronic renal or cardiovascular disease) in Period III went directly to Period VI. In Period IV participants who did not meet the blood pressure goals in Period III were randomized in a 1:2 fashion to this group or the OLM/AML/HCTZ 40/5/12.5 group.
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion. In Period IV participants who did not meet the blood pressure goals (<140/90 mm Hg; or <130/80 for participants with diabetes or chronic renal or cardiovascular disease)in Period III were randomized in a 1:2 fashion to OLM/AML/HCTZ 20/5/12.5 or this group.
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 2 tablets of hydroclororthiazide 12.5 mg. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + 2 tablets of hydroclororthiazide 12.5 mg. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- Olmesartan(OM)20mg/Amlodipine (AML)5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 20 mg/amlodipine 5 mg + two 12.5 mg hydrochlorothiazide placebo tablets. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- Olmesartan/Amlodipine 40mg/5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + two 12.5 mg hydrochlorothiazide placebo tablets. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- Olmesartan/Amlodipine 40mg/10mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + two 12.5 mg hydrochlorothiazide placebo tablets. In Periods I/II participants were randomized to this and the other 7 arms arms in a 1:1:1:1:1:1:1:1 fashion.
- OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg: In Period V responders continued on olmesartan/amlodipine/ hydrochlorothiazide 40mg/5mg/12.5 mg. A participant was considered a responder if their blood pressure was <140/90 mm Hg; <130/80 mm Hg if the participant had diabetes or chronic renal or cardiovascular disease.
- OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg; OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg: In Period V OLM/AML/HCTZ 40/5/12.5 non-responders were randomized to olmesartan/amlodipine/hydrochlorothiazide 40mg/5mg/12.5 mg or to 40mg/5mg/25 mg. A participant was considered a responder if their blood pressure was <140/90 mm Hg; <130/80 mm Hg if the participant had diabetes or chronic renal or cardiovascular disease.
- OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg: In Period V non-responders to olmesartan/amlodipine/hydrochlorothiazide 20mg/5mg/12.5 mg were up titrated to 40mg/5mg/12.5mg. A participant was considered a responder if their blood pressure was <140/90 mm Hg; <130/80 mm Hg if the participant had diabetes or chronic renal or cardiovascular disease.
- 20/5/12.5mg Responder Continued on 20/5/12.5 mg: In Period V non-responders to olmesartan/amlodipine/hydrochlorothiazide 20mg/5mg/12.5 mg continued on 20mg/5mg/12.5mg. A participant was considered a responder if their blood pressure was <140/90 mm Hg; <130/80 mm Hg if the participant had diabetes or chronic renal or cardiovascular disease.
Period: PeriodI-II (Randomized, Double-Blind)
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg | Olmesartan(OM)20mg/Amlodipine (AML)5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg | OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg | 20/5/12.5mg Responder Continued on 20/5/12.5 mg
Started | 335 | 336 | 336 | 336 | 336 | 337 | 337 | 336 | 0 | 0 | 0 | 0 | 0
Completed | 319 | 325 | 323 | 309 | 315 | 322 | 319 | 311 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 11 | 13 | 27 | 21 | 15 | 18 | 25 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 11 | 3 | 7 | 13 | 10 | 5 | 9 | 17 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 5 | 8 | 7 | 6 | 5 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 5 | 4 | 2 | 4 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Reason | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period III (Single-Blind)
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg | Olmesartan(OM)20mg/Amlodipine (AML)5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg | OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg | 20/5/12.5mg Responder Continued on 20/5/12.5 mg
Started | 2540 (2543 completed Period 2. Three decided not to continue in the study=2540.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2520 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period IV (Double-Blind)
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg | Olmesartan(OM)20mg/Amlodipine (AML)5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg | OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg | 20/5/12.5mg Responder Continued on 20/5/12.5 mg
Started | 228 (2 did not continue in the study and 1837 responders went directly to Period VI. 228+453+2+1837=2520) | 453 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 226 | 451 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period V (Double -Blind)
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg | Olmesartan(OM)20mg/Amlodipine (AML)5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg | OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg | 20/5/12.5mg Responder Continued on 20/5/12.5 mg
Started | 0 (677 completed Period 4. 1 did not continue and 2 erroneously responders were not counted = 674) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 135 | 119 | 194 | 151 | 75
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 134 | 119 | 193 | 151 | 73
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Period VI (Open-Label)
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide(HCT) 40mg/10mg/25mg | Olmesartan(OM)20mg/Amlodipine (AML)5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | OM/AML/HCT 40/5/12.5mg Responder Continued on 40/5/12.5 mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/12.5mg | OM/AML/HCT 40/5/12.5mg Non Responder Randomized to 40/5/25mg | OM/AML/HCT 20/5/12.5mg NonResponder Up Titrated to 40/5/12.5mg | 20/5/12.5mg Responder Continued on 20/5/12.5 mg
Started | 1447 (1837 from Period III+2 from Period IV + 670 from Period 5 = 2509) | 272 | 480 | 146 | 164 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 1408 | 264 | 467 | 143 | 157 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 39 | 8 | 13 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 17 | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 7 | 5 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 6 | 1 | 3 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Reason | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg | Olmesartan/Amlodipine 20mg/5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg | Total
Number analyzed (Participants) | 335 | 336 | 336 | 336 | 336 | 337 | 337 | 336 | 2689
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (10.81) | 56.8 (10.36) | 56.5 (10.92) | 57.0 (10.72) | 55.9 (11.08) | 56.1 (10.22) | 56.4 (10.4) | 57.0 (9.70) | 56.5 (10.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 171 | 184 | 181 | 178 | 185 | 170 | 192 | 1443
  Male | 153 | 165 | 152 | 155 | 158 | 152 | 167 | 144 | 1246
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  Black | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  White | 334 | 336 | 335 | 335 | 336 | 337 | 337 | 335 | 2685
Region of Enrollment [Number; unit: Participants]
  Europe | 335 | 336 | 336 | 336 | 336 | 337 | 337 | 336 | 2689

OUTCOME MEASURES:

1. Primary Outcome: Change in Seated Diastolic Blood Pressure (SeDBP).
Description: Baseline blood pressure was defined as the average values obtained at the randomization visit and at the visit prior to randomization
Time Frame: Baseline to week 10
Population: The full analysis set includes 2679 randomized patients who received at least 1 dose of double-blind medication and who provided at least one diastolic blood pressure measurement in Period I-II
Measure: Least Squares Mean (Standard Error); unit: mm HG
Groups:
- Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg: Once a day the following tablets were taken: 1 tablet of olmesartan 20 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 2 tablets of hydroclororthiazide 12.5 mg
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + 2 tablets of hydroclororthiazide 12.5 mg
- Olmesartan/Amlodipine 20mg/5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 20 mg/amlodipine 5 mg + two 12.5 mg hydrochlorothiazide placebo tablets
- Olmesartan/Amlodipine 40mg/5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + two 12.5 mg hydrochlorothiazide placebo tablets
- Olmesartan/Amlodipine 40mg/10mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 10 mg + two 12.5 mg hydrochlorothiazide placebo tablets
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg | Olmesartan/Amlodipine 20mg/5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg
Number analyzed (Participants) | 334 | 336 | 335 | 336 | 332 | 337 | 334 | 335
mm HG | -22.5 (0.48) | -22.5 (0.48) | -23.0 (0.48) | -23.9 (0.47) | -23.8 (0.48) | -20.5 (0.47) | -21.2 (0.48) | -22.1 (0.48)
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine 20mg/5mg; Test type: Superiority or Other; p = 0.0071, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p = 0.0323, ANCOVA
Statistical Analysis 3: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p = 0.0080, ANCOVA
Statistical Analysis 4: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.0071, ANCOVA
Statistical Analysis 5: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.0107, ANCOVA

2. Secondary Outcome: Change in Seated Systolic Blood Pressure (SeDBP).
Time Frame: Baseline to week 10
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg | Olmesartan/Amlodipine 20mg/5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg
Number analyzed (Participants) | 334 | 336 | 335 | 336 | 332 | 337 | 334 | 335
mm Hg | -33.2 (0.72) | -33.7 (0.72) | -35.3 (0.71) | -35.5 (0.71) | -36.2 (0.72) | -29.9 (0.71) | -30.4 (0.71) | -32.8 (0.71)
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine 20mg/5mg; Test type: Superiority or Other; p = 0.0006, ANCOVA
Statistical Analysis 2: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p = 0.0008, ANCOVA
Statistical Analysis 3: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.0034, ANCOVA
Statistical Analysis 5: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.0006, ANCOVA

3. Secondary Outcome: Number of Subjects Reaching Blood Pressure Goal at Week 10
Description: Blood pressure treatment goal was defined as blood pressure <140/90 mmHg or <130/80 mmHg for subjects with diabetes, chronic renal disease, or chronic cardiovascular disease.
Time Frame: baseline to week 10
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg | Olmesartan/Amlodipine 20mg/5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg
Number analyzed (Participants) | 334 | 336 | 335 | 336 | 332 | 337 | 334 | 335
Participants | 177 | 176 | 197 | 190 | 179 | 144 | 155 | 166
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine 20mg/5mg; Test type: Superiority or Other; p = 0.0295, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p = 0.2529, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg vs Olmesartan/Amlodipine 40mg/5mg; Test type: Superiority or Other; p = 0.0037, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.2033, Cochran-Mantel-Haenszel
Statistical Analysis 5: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg vs Olmesartan/Amlodipine 40mg/10mg; Test type: Superiority or Other; p = 0.2529, Cochran-Mantel-Haenszel

4. Secondary Outcome: Change in Seated Diastolic Blood Pressure From Week 18 to Week 22
Time Frame: Week 18 to week 22
Population: The Full Analysis Set 2=681 randomized participants who received at least 1 dose of double-blind medication and who provided at least one diastolic blood pressure measurement in Period IV
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg: Once a day the following tablets were taken: 1 tablet of olmesartan 20 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg.
  hydrochlorothiazide placebo tablet. Participants from Period III who did not meet blood pressure goals (<140/90; 130/80 for participants with diabetes, chronic renal disease, or chronic cardiovascular disease)were randomized to Period IV in a 1:2 ratio to continue olm/aml/hctz 20/5/12.5 or be up-titrated to olm/aml/hctz 40/5/12.5.
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg hydrochlorothiazide placebo tablet.
  Participants from Period III who did not meet blood pressure goals (<140/90; 130/80 for participants with diabetes, chronic renal disease, or chronic cardiovascular disease)were randomized to Period IV in a 1:2 ratio to continue olm/aml/hctz 20/5/12.5 or be up-titrated to olm/aml/hctz 40/5/12.5.
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg
Number analyzed (Participants) | 228 | 453
mm Hg | -3.3 (0.47) | -4.1 (0.37)
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg; Test type: Superiority or Other; p = 0.1135, ANCOVA

5. Secondary Outcome: Change in Seated Systolic Blood Pressure From Week 18 to Week 22
Time Frame: Week 18 to week 22
Population: The Full Analysis Set 2=681 randomized participants who received at least 1 dose of double-blind medication and who provided at least one blood pressure measurement in Period IV
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg: Once a day the following tablets were taken: 1 tablet of olmesartan 40 mg/amlodipine 5 mg + 1 tablet of hydroclororthiazide 12.5 mg + one 12.5 mg.
  hydrochlorothiazide placebo tablet. Participants from Period III who did not meet blood pressure goals (<140/90; 130/80 for participants with diabetes, chronic renal disease, or chronic cardiovascular disease)were randomized to Period IV in a 1:2 ratio to continue olm/aml/hctz 20/5/12.5 or be up-titrated to olm/aml/hctz 40/5/12.5.
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg
Number analyzed (Participants) | 228 | 453
mm Hg | -5.7 (0.71) | -6.5 (0.56)
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg; Test type: Superiority or Other; p = 0.2765, ANCOVA

6. Secondary Outcome: Number of Subjects Reaching Blood Pressure Goal From Week 18 to Week 22
Description: as for outcome 3
Time Frame: Week 18 to week 22
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg
Number analyzed (Participants) | 228 | 453
Participants | 63 | 137
Statistical Analysis 1: Comparison: Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg vs Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg; Test type: Superiority or Other; p = 0.4964, Cochran-Mantel-Haenszel

7. Secondary Outcome: Change in Seated Diastolic Blood Pressure From Week 22 to Week 26
Time Frame: Week 22 to week 26
Population: The Full Analysis Set 3=312 randomized participants who received at least one dose of double-blind medication and who provided at least one diastolic blood pressure measurement in Period V.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5: This arm contain participants who did not responded to olmesartan\amlodipine\hydrochlorothiazide 40/5/12.5 and who were randomized to that combination in Period V
- OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/25: This arm contain participants who did not respond to olmesartan\amlodipine\hydrochlorothiazide 40/5/12.5 and who were randomized to 40/5/25 in Period V
Arm/Group | OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 | OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/25
Number analyzed (Participants) | 119 | 193
mm Hg | -2.7 (0.68) | -3.8 (0.56)
Statistical Analysis 1: Comparison: OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 vs OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/25; Test type: Superiority or Other; p = 0.1301, ANCOVA
Statistical Analysis 2: Comparison: OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 vs OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/25; Test type: Superiority or Other; p = 0.01301, ANCOVA

8. Secondary Outcome: Change in Seated Systolic Blood Pressure From Week 22 to Week 26
Time Frame: Week 22 to week 26
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- OLM/AML/HCTZ40/5/12.5mg Nonresponders Randomized to 40/5/25: This arm contain participants who did not respond to olmesartan\amlodipine\hydrochlorothiazide 40/5/12.5 and who were randomized to 40/5/25 in Period V
Arm/Group | OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 | OLM/AML/HCTZ40/5/12.5mg Nonresponders Randomized to 40/5/25
Number analyzed (Participants) | 119 | 193
mm Hg | -4.5 (1.01) | -6.7 (0.84)
Statistical Analysis 1: Comparison: OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 vs OLM/AML/HCTZ40/5/12.5mg Nonresponders Randomized to 40/5/25; Test type: Superiority or Other; p = 0.0503, ANCOVA

9. Secondary Outcome: Number of Subjects Reaching Blood Pressure Goal at Week 26
Description: as for outcome 3
Time Frame: Week 22 to week 26
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/12.5 | OLM/AML/HCTZ 40/5/12.5mg Nonresponders Randomized to 40/5/25
Number analyzed (Participants) | 119 | 193
Participants | 29 | 47

10. Secondary Outcome: Change in Seated Systolic Blood Pressure (SeDBP) During Open-Label Period VI (Titration Effect From OM/AML/HCTZ 40/5/25 to 40/10/25.
Time Frame: Week 26 to week 54
Population: The number of subjects up titrated who had blood pressure values at both time points.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- OLM/AML/HCTZ 40/5/25 Titrated to 40/10/25: The participants in this arm had their study medication titrated from olmesartan\amlodipine\hydrochlorothiazide 40/5/25 to 40/10/25
Arm/Group | OLM/AML/HCTZ 40/5/25 Titrated to 40/10/25
Number analyzed (Participants) | 87
mm Hg | -11.9 (11.01)

ADVERSE EVENTS:
Time Frame: Week 1 to week 54
Description: All adverse events, whether observed by the investigator or reported by the participant were recorded on the Adverse Event electronic Case Report Form. Adverse events (AEs)were collected up to 14 days after the last study dose; for serious AEs considered to be drug related there was no time limit.
Arm/Group | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg | Olmesartan/Amlodipine 20mg/5mg | Olmesartan/Amlodipine 40mg/5mg | Olmesartan/Amlodipine 40mg/10mg
Serious Adverse Events (participants affected / at risk) | 55/329 | 9/334 | 22/331 | 3/329 | 7/332 | 1/333 | 5/332 | 7/325
Other Adverse Events (participants affected / at risk) | 12/329 | 44/334 | 13/331 | 39/329 | 45/332 | 26/333 | 38/332 | 30/325
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg (N=329) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg (N=334) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg (N=331) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg (N=329) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg (N=332) | Olmesartan/Amlodipine 20mg/5mg (N=333) | Olmesartan/Amlodipine 40mg/5mg (N=332) | Olmesartan/Amlodipine 40mg/10mg (N=325)
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QRS complex shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transient ischemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angle closure glaucoma (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Barotrauma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Removal of internal fixation (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Hepatitus B virus (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mediastinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyothorax (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abcess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vertebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0/0 | 0
Femeral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Olmesartan/Amlodipine/Hydrochlorothiazide 20mg/5mg/12.5 mg (N=329) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/12.5mg (N=334) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/5mg/25mg (N=331) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/12.5mg (N=329) | Olmesartan/Amlodipine/Hydrochlorothiazide 40mg/10mg/25mg (N=332) | Olmesartan/Amlodipine 20mg/5mg (N=333) | Olmesartan/Amlodipine 40mg/5mg (N=332) | Olmesartan/Amlodipine 40mg/10mg (N=325)
Oedema peripheral (General disorders) | 0 | 15 | 0 | 26 | 27 | 11 | 16 | 30
Headache (Nervous system disorders) | 12 | 16 | 13 | 13 | 18 | 15 | 0 | 0
Nasopharyngitis (Investigations) | 0 | 13 | 0 | 0 | 0 | 0 | 11 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A site may not publish results until after a coordinated multicentre publication has been submitted for publication or until one year after the study has ended, whichever occurs first. Then, the site will have the opportunity to publish the results, provided that DSE has had the opportunity to review and comment on the site's proposed publication prior to its being submitted for publication with the advice of company patent council and in accord with needs for subject protection.